CLINICAL TRIAL: NCT00574314
Title: Women's Health Research Registry
Status: Terminated | Type: Observational
Why Stopped: No more funding
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB# 4269; 4269
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: women; Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women: Women with varying backgrounds
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants will be consented.

SUMMARY:
Women have been disproportionately underrepresented in clinical research. Few of the many drugs approved by the FDA have been adequately tested in women. Most common health conditions experienced by both women and men are managed by treatments that have been developed and tested most in men.

A new barrier to enrolling women in clinical trials is in effect: HIPAA (the Health Insurance Portability and Accountability Act). The positive benefit of HIPAA-protecting a person's health information from abuse-is laudable, but it comes at a cost: it will deny investigators the benefit of access to chart (medical record) review in order to gather data to answer clinical questions. In the past, investigators were allowed access to patient's charts because the hospital consent form included a clause indicating that the patient's information may be used for research.

The investigators propose to overcome this crisis and challenge with a proven method of identifying individuals who would be willing to consider participating in a clinical trial: The Women's Guild Health Research Registry. In keeping with the focus of the Women's Health Program, we would propose to enroll only women. The registry will allow qualified investigators to identify potential study participants. This idea has been effective at improving the quantity and quality of women able and willing to participate in trials.

The investigators will also allow other approved sites to utilize the Registry via the approved procedure of submitting an IRB approved protocol which will be reviewed by our Internal Review Committee. This protocol's inclusion/exclusion criteria will be used to query the database for eligible participants. The participants will be contacted by the Registry staff to ascertain their interest in this research protocol and their agreement to release their contact data to the investigator will be obtained.

Investigators will be charged at the time they approach the registry for assistance. The charge is intended to cover the cost of maintaining the registry now that initial funding has been exhausted.

DETAILED DESCRIPTION:
See Brief Summary above

ELIGIBILITY:
Inclusion Criteria:

* Adult women
* English speaking

Exclusion Criteria:

* We do not include children.
* We do not include non-English speaking subjects at this time.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All adult English-speaking women
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2004-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes